CLINICAL TRIAL: NCT04525508
Title: Coronary Artery Plaque Burden in Asymptomatic Danish Men Aged 65-75 Years and the Relation to Glycemic Status. A Coronary CT Angiography (CCTA) Study.
Brief Title: Coronary Artery Plaque Burden in Asymptomatic Danish Men Aged 65-75 Years and the Relation to Glycemic Status.
Acronym: DANCAP
Status: Completed | Type: Observational
Sponsor: Svendborg Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Johanna Larsson, Johanna Larsson, Svendborg Hospital, Svendborg Hospital
Other Study IDs: 01
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease; Dysglycemia
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Storage in biobank (-80° C):
  5 x 2 ml (serum). 4 x 2 ml (ethylenediaminetetraacetic acid). 2 x 2 ml (sodium citrate)
  1 x 2 ml (erythrocyte sedimentation rate)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal glucose tolerance (NGT): Those of the study population with one normal Oral glucose tolerance test (OGTT)
- Dysglycemia: Those of the study population with one dysglycemia (IFG and/or IGT)
- Diabetic OGTT: Those of the study population with one Diabetic OGTT

SUMMARY:
Cardiovascular disease (CVD) is one of the leading causes of death in the Western Society. Patients with type 2 diabetes mellitus (T2DM) or dysglycemia have an increased risk of developing CVD. Furthermore, T2DM have an increased risk of developing heart failure, especially non-systolic, whether or not this is correlated to stepwise abnormal glycemic status is not fully investigated.

The aims of this study are to investigate association between 1) Coronary plaque burden and morphology to glycemic status (normal glucose tolerance (NGT), dysglycemia (impaired fasting glucose (IFG) or impaired glucose tolerance (IGT)) and diabetic oral glucose tolerance test (OGTT) in participants without known T2DM), 2) Coronary plaque burden and morphology to diastolic and systolic function of the left ventricle including 2D speckle-tracking assessments, 3) Glycemic status to diastolic and systolic function of the left ventricle including 2D speckle-tracking assessments

In this descriptive study, 500-800 asymptomatic men aged 65-75 without known diabetes will be included and divided into three subpopulations according to glycemic status. Blood sample, oral glucose tolerance test (OGTT), echocardiography and Coronary CT Angiography (CCTA) will be performed at inclusion

DETAILED DESCRIPTION:
Background

Cardiovascular disease: Cardiovascular disease (CVD) is still one of the leading causes of death in the Western Society. Despite extensive research, risk estimation based on traditional risk factors predicts risk in the general population but may not give an adequate individual risk, and can thereby under- or overestimate the risk of future cardiovascular event and therefore lead to either over- or undertreatment of a not ignorable part of the population.

T2DM/dysglycemia and atherosclerosis: The prevalence of type 2 diabetes mellitus (T2DM) is rising rapidly. Furthermore, one study has reported that the prevalence of dysglycemia or undiagnosed diabetes were as high as 43.8% among 60-year-old men. T2DM is known to be strongly associated with an increased risk of CVD, but also dysglycemia has been associated with an increased risk of CVD. Thus, it is possible that there is a linear relationship between stepwise dysregulated glycemic status and increased coronary plaque burden, but the relationship has not been fully explored.

CCTA: Coronary CT Angiography (CCTA) can be performed with or without contrast. Contrast enhanced CCTA has been found to be a valid and reproducible method of evaluation of both extent and characteristics of atherosclerotic plaques. Motoyama et al. reported spotty calcification, positive remodeling, and LAP (non-calcified plaque) to be associated with an increased risk of development of AMI, especially when two or more patterns were co-localized in the plaques. Thus, it might be possible that this type of plaque morphology is associated with vulnerable plaques.

Echocardiography and T2DM/Dysglycemia: T2DM is correlated to a higher incidence of diastolic dysfunction, which is thought to predispose to diabetic cardiomyopathy. In addition, subtle left ventricular systolic dysfunction assessed by 2D speckle-tracking (also termed impaired strain) was found in patients with diabetes and normal systolic function. To our knowledge only few studies have investigated diastolic dysfunction and 2D speckle-tracking in patients with dysglycemia and their results were mostly diverging.

To our knowledge no studies have investigated coronary artery plaque burden and morphology in asymptomatic men aged 65-75 years with focus on the influence of glycemic status in individuals without known T2DM. Due to the expectance of increasing number of patients with T2DM and dysglycemia the coming years, it must be foreseen that the number of patients with CVD will increase in this group of patients. It is mandatory that we increase our knowledge, especially about the development of coronary atherosclerosis and left ventricular function. We expect that this study will bring further light on these important aspects of dysglycemia and hopefully give information to improve treatment and prophylaxis.

Methods

Study population: We plan to recruit 500-800 participants from the DANCAVAS study. More detailed description of the Study population can bee read in "Eligibility". Based on one oral glucose tolerance test (OGTT) per participant, this population will be divided into three groups; normal glucose tolerance (NGT), dysglycemia (impaired fasting glucose (IFG) or impaired glucose tolerance (IGT)) and diabetic OGTT without known T2DM. We use the WHO definitions in dividing the participants into the mentioned three groups of different glycemic status. To date the use of OGTT in diagnosing T2DM, demands two measurements at two separate days. Because of the measurement of only one OGTT in this study, the participants with diabetic OGTT does not per se fulfil the criteria for diabetes.

Data acquisition

1. OGTT: Patients will be instructed in 8-12 hours fasting before the OGTT. Fasting plasma glucose (FPG) will be measured. Thereafter, 75 gram glucose will be ingested over five minutes. 120 minutes later plasma glucose (120-PG) will be measured and patients will be categorized according to mentioned definitions.
2. Echocardiography: Echocardiography standard measurements of left ventricular (LV) systolic and diastolic function:

   * LV and left atrial volumes will be estimated using Simpson's biplane method of discs in the 4 and 2-chamber views, and LV ejection fraction will be calculated.
   * The mitral inflow pattern will be estimated in the apical 4-chamber view, and the peak early (E) and peak atrial(A) velocities will be measured. Peak early mitral annular velocities (e') will be estimated using tissue Doppler imaging. The E/e´ratio will be obtained by dividing E by average value of e´.

   Global left ventricular longitudinal strain (GLS):
   * Longitudinal systolic strain will be measured using 2D speckle tracking echocardiography. This measurement will be obtained from views with an optimized focus on the LV and a frame rate of about 60-80 frames/sec. Subsequently LV will be divided into 18 segments. GLS will be calculated by the software as the mean value of the peak systolic longitudinal strain of the 18 segments.
3. CCTA: The CCTA scan GE revolution will be used. CAC score will be evaluated using non contrast scans from the DANCAVAS study. In our study, contrast enhanced scans using 256-slice, ECG-gated, will be performed. In order to regain optimal results, patients with pulse >60 beat/min will be given intravenous Beta-blockers and sublingual Nitroglycerin spray just before the examination if not contraindicated. Depending on BMI, tube voltage will be 120 or 100 kV and tube current 350-650 mAs. The collimation is 256×0,23mm with a gantry rotation time of 280 ms with 16 centimeters axial coverage per rotation. The estimated total radiation dose for one contrast enhanced CCTA is 1-6 mS. To reduce risk of contrast related affection of the kidney function a recent eGFR must be obtained before scanning and patients will be sufficiently hydrated.

   CCTA analysis:

   Plaque burden The major proximal coronary segments; 1,2,3-5,6,7-11,12,13 are analyzed.

   Per vessel analysis of:
   * Percent atheroma volume (PAV):(Total vessel volume-total lumen volume/total vessel volume×100%)
   * Total atheroma volume (TAV):(Total vessel volume-total lumen volume)
   * Normalized atheroma volume (NAV):(Total vessel volume-total lumen volume/mean segment length)

   Plaque morphology

   Per plaque analysis of:
   * LAP: defined as a non-calcified plaque (HU<150) with a lipid core of <30 HU.
   * Remolding indices (RI): calculated by lesion diameter/reference diameter, where the reference diameter is from a normal appearing proximal segment.
   * Spotty calcifications (SC): defined as small calcified nodules <3mm in length and <=90 degrees of the coronary arch.
   * Degree of stenosis: a significant stenosis is defining as >70% of the luminal area.

   All CTTA scans will be assessed by an observer blinded to patient characteristics. Semi quantitative method using dedicated plaque software (QAngioCT Research Edition version 2.0, Medis Medical Imaging Systems, Leiden, Holland) will be used to assess the plaque analysis.
4. Population characteristics: Baseline data will be collected from journal system and questionnaires and includes demographic, former CVD disease, presence of T2DM and information regarding the traditional risk factors (e.g. hypertension, hypercholesterolemia, obesity and smoking).
5. Blood sample: Blood sample includes e.g.cholesterol profile, HbA1c, Creatinine, C-Peptide, Insulin etc. Additionally, totally 30 ml blood will be collected to form a biobank for future research on the influence of inflammatory markers on atherosclerosis and glycemic status.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 years
* Capable of giving written informed consent
* Participates in the DANCAVAS study

Exclusion Criteria:

* Body mass index (BMI) >35
* Atrial fibrillation and other tachyarrhythmia that unable CCTA analysis
* Estimates Glomerular filtration rate (eGFR) <45 ml/min
* Contrast allergy
* Untreated hyperthyroid
* History of CAD or Apoplexia
* Symptoms of CAD
* Known Diabetes Mellitus

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: We will recruit participants from the DANCAVAS study. The DANCAVAS study will include 45.000 men aged 65-74 years. 15.000 of the participants will be randomly selected to CCTA (non-contrast) and the resulting 30.000 constitutes the control group. The CCTA will be performed in four Danish cities. Our study will include 500-800 of those DANCAVAS participants who will undergo CCTA in OUH Svendborg Hospital. In our study we will perform following examination in addition to the examinations in the DANCAVAS study: one CCTA (contrast enhanched), one echocardiography and one OGTT.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2016-05; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Correlation between glycemic status to coronary plaque burden and morphology. | Baseline
  To evaluate the correlation between glycemic status (NGT, dysglycemia or Diabetic OGTT in patients without known T2DM) to plaque burden and morphology in asymptomatic men, aged 65-75 years. Plaque burden analyzed per vessel is defined as either percent atheroma volume (PAV), total atheroma volume (TAV) or normalized atheroma volume (NAV). Plaque morphology will include per plaque analysis of LAP (noncalcified plaque), remodeling indices (RI), spotty calcification and degree of stenosis where a significant stenosis is defined as >70 % of the luminal area. Above mentioned definitions of plaque burden and morphology is further explained in detail in Study Description above.

SECONDARY OUTCOMES:
Association between coronary artery plaque burden and morphology to diastolic and systolic function of the left ventricle. | Baseline
  To evaluate the correlation between coronary artery plaque burden and morphology to diastolic and systolic function of the left ventricle in asymptomatic men, aged 65-75 years without known T2DM. We will use EF and 2D speckle-tracking to asses the systolic function of the left ventricle.
Association between glycemic status to diastolic and systolic function of the left ventricle. | Baseline
  To evaluate the correlation between glycemic status to diastolic and systolic function of the left ventricle in a population of asymptomatic men, aged 65-75 years without known T2DM.

OTHER OUTCOMES:
Association between insulin resistance to coronary artery plaque burden and morphology. | Baseline
  To evaluate the possible association between insulin resistance to coronary artery plaque burden and morphology in asymptomatic men, age 65-75 years without known T2DM. We will use HOMA-IR to asses the insulin resistance.
Correlation between insulin resistance to diastolic and systolic function of the left ventricle. | Baseline
  To evaluate the relation between insulin resistance to diastolic and systolic function of the left ventricle in asymptomatic men, aged 65-75 years without known T2DM.
Correlation between inflammatory biomarkers eg. TNF-alpha and Hs-CRP to coronary artery plaque burden and morphology. | Baseline
  To evaluate the correlation between inflammatory biomarkers eg. TNF-alpha and Hs-CRP to coronary artery plaque burden and morphology in a population consisting of asymptomatic men, aged 65-75 years, without known T2DM.
Association between glycemic status to left ventricular hypertrophy. | Baseline
  To evaluate the association between glycemic status to left ventricular hypertrophy in asymptomatic men, aged 65-75 years, without known T2DM.
Correlation between risk factors for ischemic heart disease to coronary artery plaque burden and morphology. | Baseline
  To evaluate the correlation between risk factors for ischemic heart disease to coronary artery plaque burden and morphology in asymptomatic men, aged 65-75 years, without known T2DM
Correlation between plaque burden and morphology to future cardiovascular events. | Baseline - 5 years
  To evaluate the correlation between plaque burden and morphology to future cardiovascular events during five years of follow up, in a population of asymptomatic men aged 65-75 years without known T2DM.
Impact of glycemic status to future cardiovascular events. | Baseline - 5 years
  To evaluate the impact of glycemic status to future cardiovascular events during five years of follow up, in a population of asymptomatic men aged 65-75 years without known T2DM.
Association between coronary plaque burden and morphology to post-systolic shortening. | Baseline
  To evaluate the impact of coronary plaque burden and morphology to post-systolic shortening in asymptomatic men, aged 65-75 years without known T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Larsson, MD, Principal Investigator — Svendborg Hospital
Locations (1):
- Cardiovascular Research Unit, OUH Svendborg Hospital, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No